CLINICAL TRIAL: NCT07281755
Title: Objective Mobility Assessment Using Wearable Technology for Clinical Application in Parkinson's Disease: From Validation to Fall Prediction
Status: Recruiting | Type: Observational
Sponsor: Northumbria University (Other)
Collaborators: DANU Sports Ltd (Unknown)
Responsible Party: Principal Investigator, GabriellaGatti, Postgraduate Researcher, Northumbria University
Other Study IDs: 8543a
Record Dates: First submitted 2025-09-16; First posted 2025-12-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease(PD)
Keywords: DANU; Wearable Electronic Devices; Gait Analysis; Validity and Reliability; Mobility Assessment; Smart Socks
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's Disease (PD): People with a clinical diagnosis of Parkinson's Disease will be recruited to participate within the study. All participants must fit within the described eligibility criteria.
  Within the verification and analytical validation phase 30 people with Parkinson's will be recruited and within clinical validation 60 individuals will be recruited.

SUMMARY:
The main objective of this observational trial is to explore the validity and reliability of DANU smart socks when used for mobility assessments in people with Parkinson's. Using a series of laboratory gold standard equipment, this project aims to compare the metrics observed by DANU to the reference standards. No intervention is included. Specifically, this study will explore metrics relating to walking (gait) and balance of a Parkinson's cohort through a series of motor tasks. Moreover, this study seeks to investigate the clinical validity of DANU outcome metrics exploring relationships with clinical scales, fall history and prospective falls.

DETAILED DESCRIPTION:
Background:

Mobility impairments are common in Parkinson's disease (PD) and increase the risk of falling. Data derived from wearable inertial measurement units can provide useful information regarding gait in different situations and environments, which may help to identify those at risk of falling. However, rigorous testing is required to evaluate whether new devices are fit for purpose. DANU Smart Socks are a multi-modal system for movement analysis, containing 15 silicone based capacitive pressure sensors and an IMU pod, with tri-axal accelerometers, gyroscope and magnetometers, currently at use within a sporting context. Potential has been highlighted for clinical use in people with Parkinson's (PwP). This study aims to evaluate the validity, reliability and usability of the DANU Sport System in PwP for balance and gait assessment. The V3+ framework for determining fit-for-purpose biometric monitoring devices will be employed, evaluating verification, usability, analytical and clinical validation.

Methods:

Institutional ethics have been obtained (Project ID: 8543). Utilising a a repeated measures observational design, participants will be asked to attend two visits to Northumbria University, Newcastle Upon Tyne.

Visit 1: Participants will complete a series of clinical and cognitive measures including the Movement Disorders Society's-Unified Parkinson's Disease Rating Scale, Montreal Cognitive Assessment, Freezing of Gait Questionnaire and Falls Efficacy Scale. Following this, concurrent data collection will occur throughout a battery of motor tasks to observe gait/balance metrics. Laboratory references employed include Axivity AX6, Vicon 3D Motion Capture, APDM Mobility Lab, GAITRite and AMTI Force Plates. Mobility assessments include a 2-Minute Walk Test, 3 walkway trials, a Timed Up and Go and a series of 2-Minute Balance tasks.

Visit 2: Participants attend a second visit to repeat the mobility assessment previously detailed utilizing DANU Smart Socks and APDM Mobility Lab systems to explore test-retest reliability.

Wearable device (DANU) validity and reliability will be examined using intra-class correlation coefficients and Bland-Altman plots to compare to laboratory reference standards. Moreover time series plots will be employed to evaluate the raw data agreement.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's by a movement disorder specialist according to UK brain bank criteria.
* Hoehn & Yahr stages I-III
* Able to attend Northumbria University, Newcastle Upon Tyne for study visits
* Able to walk and stand unassisted for a minimum of 2-minutes

Exclusion Criteria:

* History of neurological disorders other than PD (e.g., Huntington's disease, stroke, traumatic brain injury, multiple sclerosis, Alzheimer's disease etc.)
* Montreal Cognitive Assessment (MoCA) score < 21
* Injury to the lower extremities within the past 6-weeks.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Within laboratory testing, 60 people with Parkinson's (H&Y I-III) are aimed to be recruited from the North East region of England.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Stride Length | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (m, mean ± standard deviation)
Step Time | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (s, mean ± standard deviation)
Stride Time | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (s, mean ± standard deviation)
Cadence | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (steps per minute, mean ± standard deviation)
Ground Contact Time | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (s, mean ± standard deviation)
Swing Time | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (s, mean ± standard deviation)
Stride Velocity | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (m/s, mean ± standard deviation)
Gait Velocity | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (m/s, mean ± standard deviation)
Area of Ellipse | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (mm², mean ± standard deviation)
Length of Ellipse | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (mm, mean ± standard deviation)
Width of Ellipse | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (mm, mean ± standard deviation)
Total Displacement | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (mm, mean ± standard deviation)
Medio-Lateral Range | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (mm, mean ± standard deviation)
Anterior-Posterior Range | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (mm, mean ± standard deviation)

OTHER OUTCOMES:
Double Support Time | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (s, mean ± standard deviation)
Single Support Time | Outcomes will be obtained on Visit 1 (Day 1) and Visit 2 (Day 8).
  (s, mean ± standard deviation)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Vitorio, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: DANU Medical Website: Study Collaborator and Smart Sock System. — https://www.danumedical.com/